CLINICAL TRIAL: NCT03487471
Title: Comparison of Accuracy and Reproducibility of Breast Lesion Characterization Between Real Time Elastography and Shear Wave Elastography
Brief Title: Comparison of Real-time and Shear Wave Elastography
Acronym: Elasto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Elasto Trial
Record Dates: First submitted 2018-03-16; First posted 2018-04-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time elastography (Active Comparator): 98 patients with breast lesion will a receive breast ultrasound (real time elastography)
  Interventions: Diagnostic Test: Real-time elastography
- Shear Wave (Active Comparator): 98 patients with breast lesion will a receive breast ultrasound (shear wave elastography)
  Interventions: Diagnostic Test: Shear wave elastography

INTERVENTIONS:
Diagnostic Test: Real-time elastography — Breast ultrasound with real-time elastography
  Arms: Real-time elastography
Diagnostic Test: Shear wave elastography — Breast ultrasound with shear wave elastography
  Arms: Shear Wave

SUMMARY:
Tissue elasticity is being increasingly used as diagnostic parameter, since at the macroscopic level benign breast lesions tend to be stiffer than normal breast tissue but softer than breast cancers. Ultrasound elastography allows to probe the elasticity of breast lesions in clinics. Real time elastography (RTE) and shear wave elastography (SWE) are the two most widely used elastography modalities.

Assessment of breast lesions by either RTE or SWE improve the diagnostic performance of standard B-mode ultrasound (US) and have the potential to assist the decision about whether to perform a breast biopsy or not.

DETAILED DESCRIPTION:
Tissue elasticity is being increasingly used as diagnostic parameter, since at the macroscopic level benign breast lesions tend to be stiffer than normal breast tissue but softer than breast cancers. Ultrasound elastography allows to probe the elasticity of breast lesions in clinics. Real time elastography (RTE) and shear wave elastography (SWE) are the two most widely used elastography modalities.

Assessment of breast lesions by either RTE or SWE improve the diagnostic performance of standard B-mode ultrasound (US) and have the potential to assist the decision about whether to perform a breast biopsy or not. However, employing RTE and SWE using the same equipment to directly compare elasticity measurements of a breast lesion has not been done. Investigators propose to prospectively investigate inter-observer agreement of each modality.

The study will investigate and compare the accuracy and reproducibility of SWE and RTE in the characterization of breast lesions. Furthermore, we plan to establish learning curves for RTE and SWE.

In this project, investigators will compare RTE and SWE concerning their potential to discriminate benign breast lesions from breast cancer. Investigators aim is to identify which modality will allow clinicians the best possible patient care.

ELIGIBILITY:
Inclusion Criteria:

* Female patients at least 18 years of age with a known breast lesion
* Signed informed consent

Exclusion Criteria:

* Male
* Younger than 18 years of age
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 98 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
assessment of dignity of breast lesion by use of real-time elastography | at baseline
  variability in breast lesion diagnostics by use of real-time elastography versus shear wave elastography
assessment of dignity of breast lesion by use of shear wave elastography | at baseline
  variability in breast lesion diagnostics by use of real-time elastography versus shear wave elastography

SECONDARY OUTCOMES:
Examinators learning curve | baseline until year 1
  Establish learning curves for real-time elastography and shear wave elastography

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Zanetti, Principal Investigator — St Claraspital Basel
Locations (1):
- St Claraspital, Basel, Switzerland